CLINICAL TRIAL: NCT05024981
Title: Videographic Feedback and Walk Rehabilitation in Post-Cerebrovascular Accident
Acronym: CoDévi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-GIRCI-02
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Classic reeducation (Active Comparator)
  Interventions: Behavioral: Classic reeducation
- Classic reeducation + videographic feedback (Experimental)
  Interventions: Behavioral: Videographic feedback

INTERVENTIONS:
Behavioral: Videographic feedback — Twice a week during his classic re-education sessions, the patient will be filmed for 1 minute. After transferring the video to a tablet, he will watch the video once and decide what he wants to correct. During the second viewing, he will analyse his walk, the therapist being present to provide additional information. Finally, the patient will apply his analysis while being filmed and will compare the possible differences between the 2 videos. Depending on the time available, the patient may have to repeat the recordings, analyses and exercises.
  Arms: Classic reeducation + videographic feedback
Behavioral: Classic reeducation — The patient will benefit twice a day for 30 minutes from re-education sessions.
  Arms: Classic reeducation

SUMMARY:
Cerebrovascular Accident affects the majority of the elderly population and its frequency is constantly increasing. The resulting deficits are numerous and lead in particular to an alteration in the quality of walking and autonomy. Numerous rehabilitation techniques have been described. In practice, correction instructions are often given by the therapist while the motor activity is being performed. Walking is a complex activity, as is the processing of dual-task information in elderly stroke patients. It therefore appears interesting to separate the time of motor realization and that of correction instructions. Investigators therefore propose firstly to film the patient during the performance of a walking activity and then, secondly, to analyse the video with the patient, which thus represents a source of delayed feedback. The main objective of the study is to observe the effects of this practice on walking speed. Investigators are comparing two groups of patients: the control group receiving conventional rehabilitation and the experimental group receiving conventional rehabilitation plus sessions with the video tool. They expect to observe a greater improvement in walking speed in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for a first episode of Cerebrovascular Accident less than six months old, or nth stroke less than six months old, with no previous sequelae;
* Able to walk at least 10m without stopping, with or without technical assistance, but without human assistance, under supervision;

Exclusion Criteria:

* Palliative or life-threatening situation;
* A patient whose guardian or trustee is not readily available to provide information about the patient
* Neuro-cognitive disorder that prevents understanding of instructions, as determined by the clinician;
* Severe speech or language disorder that prevents the protocol from being carried out correctly;
* Hemineglect;
* Any previously known pathology altering the gait pattern, at the clinician's discretion (recent neurological, traumatological or orthopaedic pathologies, etc.);
* Visual disorder preventing viewing of the video;
* Hearing disorder preventing comprehension.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Day 26
  Difference in walking speed between the initial and final assessment in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey MARTEU, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU Nice, Nice, Alpes-Maritime, France

IPD SHARING:
Plan to Share IPD: No